CLINICAL TRIAL: NCT03434626
Title: A Randomized Trial of ACP/GCD Care Pathway in Primary Care in Alberta
Brief Title: Advance Care Planning & Goals of Care Randomized Controlled Trial in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Queen's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 06-17
Record Dates: First submitted 2017-08-01; First posted 2018-02-15 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Chronic Illness; Comorbidities
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor conducting interviews does not have information on group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACP Education (Experimental): Eligible patients in the experimental group will receive an educational intervention from an advance care planning navigator consisting of a 4-item values tool, a Goals of Care Designation form and, if applicable, watch a cardiopulmonary resuscitation video.
  Interventions: Behavioral: ACP Education; Other: Usual care
- Usual care (Active Comparator): Patients in the usual care group will complete a Goals of Care Designation form with the family physician.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: ACP Education — Decision aid and Goals of Care Designation form information administered by Navigator
  Arms: ACP Education
Other: Usual care — Usual care includes reviewing Goals of Care Designation form and Greensleeve with physician

SUMMARY:
Sometimes people with health conditions become ill suddenly and can no longer speak for themselves and another person (such as a family member) will make health care decisions for them. This means it is important for people to think about their wishes and tell others about them. This is called advance care planning. When people have done advance care planning, if they become very sick and cannot speak for themselves they are more likely to get the kind of health care they want and it is easier for the people who make decisions for them. In Alberta, there is a form in the health care system that is used to indicate a person's wishes if participants are unable to speak for themselves. There are tools such as brochures, questionnaires, and videos that can help participants learn about advance care planning and serious illness conversations. This research is being done to study whether using tools for advance care planning will help improve goals of care designation completion rates in such a way that they better reflect patient values. In this project, we aim to determine the efficacy of tools to increase the quality and quantity of advance care planning (ACP) and Goals of Care Determinations (GCD) in primary care settings in Alberta.

DETAILED DESCRIPTION:
In prospective and randomized trials, advance care planning (ACP) significantly improves outcomes including increased likelihood that clinicians and families understand and comply with a patient's wishes, reduces hospitalization at the end of life, results in less intensive treatments at the end of life (according to patients' wishes) and increases use of hospice services. Trials have not been done in primary care. The aim of this study is to determine the efficacy of a care pathway designed to increase the quality and quantity of ACP in patients and their substitute decision-makers in primary care. The study is a multi-site, patient-based, unblinded, randomized trial conducted in family practices in Canada. Participants will be patients who are determined by their physician to be able to benefit from ACP, and the patient's substitute decision-maker. Participant pairs will be randomized to immediate intervention (care pathway) or delayed (8-12 weeks). The intervention is guided use of tools and decision aids to clarify values and preferences for treatments in the event of serious illness or near end of life. The outcomes will be presence of a goals of care form in the chart, substitute decision-maker engagement in ACP (including self-efficacy for enacting the role), patient engagement in ACP, and decisional conflict.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* have at least one chronic condition that may be life-limiting

Exclusion Criteria:

* Unable to communicate with an English-speaking research coordinator

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Presence of a completed goals of care designation form in the patient chart | 8-12 weeks
  In Alberta there is a form in the health care system that is used to indicate a person's wishes if they are unable to speak for themselves. The form is called a "Goal of Care Designation" form and is part of a package called the 'Greensleeve'. Alberta Health Services requires that all patients in primary care and in hospital have a green sleeve and goal of care designation (RMC classification: R=resuscitative; M=medical; C=comfort care).

SECONDARY OUTCOMES:
Agreement between patient's self-reported values and preferences for life sustaining treatment, and what is documented in the form in the chart | 8-12 weeks
  Dichotomous variable of whether there is concordance between what the patient reports and what is in their chart (difference between groups)
Physician rating of decisional conflict | 8-12 weeks
  The decisional conflict scale (DCS) measures personal perceptions of uncertainty in choosing options;modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and effective decision making. The outcome is the agreement between patient's self-reported preference for life sustaining treatment and decisional conflict using a 5-item decisional conflict scale pre- and post-intervention. Each item is scored 0 to 4 (0=Yes; 1=Probably Yes; 2=Unsure; 3=Probably No; 4=No)
Patient-reported satisfaction with the intervention | 8-12 weeks
  Do patients who participate in an ACP educational intervention experience greater satisfaction with decision-making than patients who get usual care?

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Howard, PHD, Principal Investigator — McMaster University; Daren K Heyland, MD, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Family Medical Centre, Lethbridge, Alberta
  - Chinook Primary Care Network, Lethbridge, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ehlenbach WJ, Barnato AE, Curtis JR, Kreuter W, Koepsell TD, Deyo RA, Stapleton RD. Epidemiologic study of in-hospital cardiopulmonary resuscitation in the elderly. N Engl J Med. 2009 Jul 2;361(1):22-31. doi: 10.1056/NEJMoa0810245. PMID 19571280
- [Result] Heyland DK, Lavery JV, Tranmer JE, Shortt SE, Taylor SJ. Dying in Canada: is it an institutionalized, technologically supported experience? J Palliat Care. 2000 Oct;16 Suppl:S10-6. PMID 11075528
- [Result] Gruneir A, Mor V, Weitzen S, Truchil R, Teno J, Roy J. Where people die: a multilevel approach to understanding influences on site of death in America. Med Care Res Rev. 2007 Aug;64(4):351-78. doi: 10.1177/1077558707301810. PMID 17684107
- [Result] Cook D, Rocker G, Marshall J, Sjokvist P, Dodek P, Griffith L, Freitag A, Varon J, Bradley C, Levy M, Finfer S, Hamielec C, McMullin J, Weaver B, Walter S, Guyatt G; Level of Care Study Investigators and the Canadian Critical Care Trials Group. Withdrawal of mechanical ventilation in anticipation of death in the intensive care unit. N Engl J Med. 2003 Sep 18;349(12):1123-32. doi: 10.1056/NEJMoa030083. PMID 13679526
- [Result] Heyland DK, Barwich D, Pichora D, Dodek P, Lamontagne F, You JJ, Tayler C, Porterfield P, Sinuff T, Simon J; ACCEPT (Advance Care Planning Evaluation in Elderly Patients) Study Team; Canadian Researchers at the End of Life Network (CARENET). Failure to engage hospitalized elderly patients and their families in advance care planning. JAMA Intern Med. 2013 May 13;173(9):778-87. doi: 10.1001/jamainternmed.2013.180. PMID 23545563
- [Result] You JJ, Dodek P, Lamontagne F, Downar J, Sinuff T, Jiang X, Day AG, Heyland DK; ACCEPT Study Team and the Canadian Researchers at the End of Life Network (CARENET). What really matters in end-of-life discussions? Perspectives of patients in hospital with serious illness and their families. CMAJ. 2014 Dec 9;186(18):E679-87. doi: 10.1503/cmaj.140673. Epub 2014 Nov 3. PMID 25367427
- [Result] Heyland DK, Ilan R, Jiang X, You JJ, Dodek P. The prevalence of medical error related to end-of-life communication in Canadian hospitals: results of a multicentre observational study. BMJ Qual Saf. 2016 Sep;25(9):671-9. doi: 10.1136/bmjqs-2015-004567. Epub 2015 Nov 9. PMID 26554026
- [Result] Fried TR, Redding CA, Robbins ML, O'Leary JR, Iannone L. Agreement between older persons and their surrogate decision-makers regarding participation in advance care planning. J Am Geriatr Soc. 2011 Jun;59(6):1105-9. doi: 10.1111/j.1532-5415.2011.03412.x. Epub 2011 Jun 7. PMID 21649619
- [Result] Raymont V, Bingley W, Buchanan A, David AS, Hayward P, Wessely S, Hotopf M. Prevalence of mental incapacity in medical inpatients and associated risk factors: cross-sectional study. Lancet. 2004 Oct 16-22;364(9443):1421-7. doi: 10.1016/S0140-6736(04)17224-3. PMID 15488217
- [Result] Silveira MJ, Kim SY, Langa KM. Advance directives and outcomes of surrogate decision making before death. N Engl J Med. 2010 Apr 1;362(13):1211-8. doi: 10.1056/NEJMsa0907901. PMID 20357283
- [Result] Hammes BJ, Rooney BL. Death and end-of-life planning in one midwestern community. Arch Intern Med. 1998 Feb 23;158(4):383-90. doi: 10.1001/archinte.158.4.383. PMID 9487236
- [Result] Detering KM, Hancock AD, Reade MC, Silvester W. The impact of advance care planning on end of life care in elderly patients: randomised controlled trial. BMJ. 2010 Mar 23;340:c1345. doi: 10.1136/bmj.c1345. PMID 20332506
- [Result] Teno JM, Fisher ES, Hamel MB, Coppola K, Dawson NV. Medical care inconsistent with patients' treatment goals: association with 1-year Medicare resource use and survival. J Am Geriatr Soc. 2002 Mar;50(3):496-500. doi: 10.1046/j.1532-5415.2002.50116.x. PMID 11943046
- [Result] Houben CHM, Spruit MA, Groenen MTJ, Wouters EFM, Janssen DJA. Efficacy of advance care planning: a systematic review and meta-analysis. J Am Med Dir Assoc. 2014 Jul;15(7):477-489. doi: 10.1016/j.jamda.2014.01.008. Epub 2014 Mar 2. PMID 24598477
- [Result] Sudore RL, Lum HD, You JJ, Hanson LC, Meier DE, Pantilat SZ, Matlock DD, Rietjens JAC, Korfage IJ, Ritchie CS, Kutner JS, Teno JM, Thomas J, McMahan RD, Heyland DK. Defining Advance Care Planning for Adults: A Consensus Definition From a Multidisciplinary Delphi Panel. J Pain Symptom Manage. 2017 May;53(5):821-832.e1. doi: 10.1016/j.jpainsymman.2016.12.331. Epub 2017 Jan 3. PMID 28062339
- [Result] Robinson C, Kolesar S, Boyko M, Berkowitz J, Calam B, Collins M. Awareness of do-not-resuscitate orders: what do patients know and want? Can Fam Physician. 2012 Apr;58(4):e229-33. PMID 22611610
- [Result] Rhee JJ, Zwar NA, Kemp LA. Advance care planning and interpersonal relationships: a two-way street. Fam Pract. 2013 Apr;30(2):219-26. doi: 10.1093/fampra/cms063. Epub 2012 Oct 1. PMID 23028000
- [Result] Howard M, Bernard C, Tan A, Slaven M, Klein D, Heyland DK. Advance care planning: Let's start sooner. Can Fam Physician. 2015 Aug;61(8):663-5. No abstract available. PMID 26273075
- [Result] Teixeira AA, Hanvey L, Tayler C, Barwich D, Baxter S, Heyland DK; Canadian Researchers at End of Life Network (CARENET). What do Canadians think of advanced care planning? Findings from an online opinion poll. BMJ Support Palliat Care. 2015 Mar;5(1):40-7. doi: 10.1136/bmjspcare-2013-000473. Epub 2013 Oct 4. PMID 24644188
- [Result] De Vleminck A, Houttekier D, Pardon K, Deschepper R, Van Audenhove C, Vander Stichele R, Deliens L. Barriers and facilitators for general practitioners to engage in advance care planning: a systematic review. Scand J Prim Health Care. 2013 Dec;31(4):215-26. doi: 10.3109/02813432.2013.854590. PMID 24299046
- [Result] Johnston SC, Pfeifer MP, McNutt R. The discussion about advance directives. Patient and physician opinions regarding when and how it should be conducted. End of Life Study Group. Arch Intern Med. 1995 May 22;155(10):1025-30. doi: 10.1001/archinte.155.10.1025. PMID 7748044